CLINICAL TRIAL: NCT03745482
Title: The Impact of Unilateral Lumbar Mobilisations on Hamstring Strength, sEMG Activity and Failure Point of the Hamstring Nordic Exercise
Brief Title: The Impact of Unilateral Lumbar Mobilisations on Hamstring Strength and Failure Point of the Hamstring Nordic Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Teesside University (Other)
Responsible Party: Principal Investigator, Paul Chesterton, Senior Lecturer Sport and Exercise, Teesside University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TeessideUniversity
Record Dates: First submitted 2018-11-14; First posted 2018-11-19 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Hamstring Injury

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobilisations (Experimental): The intervention will consist of unilateral lumbar mobilisations at the L4 and L5 level in a Posterior Anterior direction. The plinth will rest on force plates to allow the authors to analyse the force placed through the vertebrae. Grade three mobilisations will be applied for a one minute period three times at both L4 and L5 level. Each level will be determined by a passive physiological intervertebral movement. Participants will receive the mobilisations at L5 first for one minute followed by L4. This is an appropriate dose for mobilisation application (Maitland, 2013). This process will be carried out three times.
  Following application of the mobilisations outcome measures including hamstring strength, sEMG activity and 3D motion analysis will take place.
  Interventions: Other: Lumbar Mobilisations
- Control (No Intervention): The control condition will consist of the participant lying prone on a plinth for the same time if takes for intervention to be applied approximately 10 minutes.
  Following the control condition outcome measures including hamstring strength, sEMG activity and 3D motion analysis will take place.

INTERVENTIONS:
Other: Lumbar Mobilisations — The intervention will consist of unilateral lumbar mobilisations at the L4 and L5 level in a Posterior Anterior direction. The side of the mobilisation will be determined by dominant leg - considered the kicking foot. The mobilisations will be administered by a physiotherapist with at least 10 years clinical experience. Teksan grip sensors will be worn by the physiotherapist to calculate the force applied to the participant. Grade three mobilisations will be applied for a one minute period three times at both L4 and L5 level. Each level will be determined by a passive physiological intervertebral movement. Participants will receive the mobilisations at L5 first for one minute followed by L4. This is an appropriate dose for mobilisation application (Maitland, 2013). This process will be carried out three times.
  Arms: Mobilisations

SUMMARY:
The aim of this study is to build on previous published work, which has indicated lumbar mobilisations have the ability to increase hamstring extensibility and decrease muscle activity. The primary aim of this project is investigate if lumbar mobilisations have an affect on the Nordic Hamstring exercise.

Aim: To investigate the short-term effects L4 and L5 Unilateral Posterior Anterior (UPA) Mobilisations on the lumbar spine on the Nordic Hamstring Exercise. Measures will include hamstring peak torque, sEMG activity and knee angle at first rapid change in angular acceleration.

DETAILED DESCRIPTION:
The study aims to investigate the short-term effects L4 and L5 Unilateral Posterior Anterior (UPA) Mobilisations on the lumbar spine on the Nordic Hamstring Exercise. Measures will include hamstring peak torque, sEMG activity and knee angle at first rapid change in angular acceleration.

Recruitment will take place via flyer and email. All testing will take place in the biodex laboratory at Teesside University. Due to the nature of the cross-over design participants will attend the laboratory six times, two for familiarisation sessions, and a remaining four testing session all 72 hours apart. The four testing sessions will contain two control and two intervention sessions attended in a randomised order.

Following recruitment participants will be required to complete a medical questionnaire and sign a consent form following reading the participant information sheet.

The Nordic Hamstring exercise will be performed by each participant across the intervention and control conditions. Participants will watch a video of a subject completing the Nordic exercise program. They will also receive the following verbal instructions:

'Players start in a kneeling position, with the torso from the knees upward held rigid and straight. The training partner ensures that the player's feet are in contact with the ground throughout the exercise by applying pressure to the player's heels/lower legs. The player then lowers his upper body to the ground, as slowly as possible to maximize loading in the eccentric phase. Hands and arms are used to break his forward fall and to push him back up after the chest has touched the ground, to minimize loading in the concentric phase (Mjølsne et al, 2005; Petersen et al, 2011).

All participants will be given the opportunity to ask questions as necessary.

A standardised warm-up on an ergometer will be undertaken for 5 minutes at 60% max resting heart rate.

Following the warm-up all participants will familiarise themselves with the Nordic Hamstring Exercise on the hamstring solo equipment. They will be able to practice up to 8 repetitions. This data will be used for a reliability study to understand the number of required repetitions for the main study.

During testing participants will attend the same laboratory for the remaining four testing sessions. They will receive two intervention sessions, when the lumbar mobilisations will be performed, and two when the control is administered.

The same warm-up undertaken during the familiarisation session will be undertaken prior to testing.

The intervention will consist of unilateral lumbar mobilisations at the L4 and L5 level in a Posterior Anterior direction. The side of the mobilisation will be determined by dominate leg - considered the kicking foot. The mobilisations will be administered by a physiotherapist with at least 12 years clinical experience. Teksan grip sensors will be worn by the physiotherapist to calculate the force applied to the participant. Grade three mobilisations will be applied for a one minute period three times at both L4 and L5 level.

For the control, all participants will be laid prone on the medical plinth in the same position will no mobilisations administered.

Outcome measures will include collection of hamstring peak force data, sEMG of the Biceps Femoris, 3D Motion capture data and subjective likert scale of exercise difficulty.

ELIGIBILITY:
Inclusion Criteria:

Current Teesside University Students/Staff 18+ years Engaged in Football related activity once a week Provide Informed Consent No current musculoskeletal Injury

Exclusion Criteria:

Current symptomatic low back pain or lower limb pathology including any injuries to the lower limb/lumbar spine within the last 6 months Previous ACL/Hamstring Rupture tear or diagnosed anterior knee pain. Under supervision of another health clinician Medical questionnaire not completed Red flags on medical questionnaire Any neurological problems Contraindications or precautions to spinal mobilisation

* malignancy, inflammatory or infectious processes involving the spine or peripheral joints,
* osteoporosis,
* spinal disorders including spondylolisthesis, ankylosing spondylitis, spinal fusion

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2019-01-04 (Actual); Primary Completion 2019-09-08 (Actual); Study Completion 2020-01-10 (Actual)

PRIMARY OUTCOMES:
Hamstring Peak Force | Immediate data collection during Nordic Hamstring Exercise
  Peak Force of the Hamstring as measured by the Hamstring Solo Device during a Nordic eccentric hamstring exercise The hamstring solo device calculates Force (N), time of exercise (secs), Torque (Nm) and Torque per kg. This is collected in real-time.
  The hamstring solo calculates the eccentric force of the hamstring in real time. Participants are placed on the board with their ankle strapped. They follow previously discussed instructions to eccentrically lower themselves to the ground from a kneeling position.
sEMG of Biceps Femoris | Immediate data collection during Nordic Hamstring Exercise
  Record electromyography (SEMG) activity in the muscles of the participants in this study the Zerowire Cometa system will be used. Every electrode unit is equipped with a small unit for signal processing and transmission to the data receiver. The electrodes are single use disposable, self-adhesive silver chloride dual snap on electrodes pre-set at a distance of 20mm. All participants will have the skin prepared prior to the noraxon electrode being placed on their skin. Electrodes will be attached according to European recommendation (seniam) to the Biceps Femoris of both limbs. The electrode placement and sEMG recording will be taken by a qualified laboratory technician employed by Teesside University.
Vicon 3D Motion Capture | Immediate data collection during Nordic Hamstring Exercise
  Participants will have their mass (kg), height (cm), knee joint (between the medial and lateral epicondyle), ankle joint width (malleoli) and leg length (ASIS to medial malleolus) measured prior to recording.Widths will be measured using anthropometric calipers. Stretch height will be performed to improve the accuracy of the measurement.
  Six wall-mounted Vicon MX13 infrared cameras (Vicon) will collect 3D motion capture data at a sampling frequency of 100 Hz.. 3D motion capture data will be processed via Vicon Nexus version 1.8.5 using inbuilt pipeline functions to calculate 3D kinematic data (hip,pelvis, knee). Participants will have retroflective markers (14 mm) attached to the following landmarks on both the right and left side of the body; ASIS, PSIS, greater trochanter, mid-thigh, lateral epicondyle (of the knee), mid-tibia, lateral malleolus, calcaneus, and 2nd toe. The markers will be affixed with double-sided tape placed on the overlaying skin of the bony landmark.

SECONDARY OUTCOMES:
Subjective Likert Scale | Immediate post Nordic hamstring Exercise
  Following the Nordic exercise participants will be asked to rate the difficulty of the exercise on a 0-10 likert scale.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Chesterton, MSc, Principal Investigator — Teesside University
Locations (1):
- School of Social Sciences, Humanities and Law, Middlesbrough, Tyne and Wear, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Chesterton P, Payton S, McLaren S. Acute effects of centrally- and unilaterally-applied posterior-anterior mobilizations of the lumbar spine on lumbar range of motion, hamstring extensibility and muscle activation. J Back Musculoskelet Rehabil. 2018;31(6):1013-1023. doi: 10.3233/BMR-171000. PMID 30347590
- [Result] Chesterton P & Payton S (2017) Effects of spinal mobilisations on lumbar and hamstring ROM and sEMG: A randomised control trial. Physiotherapy Practice and Research, 38, 17-25